CLINICAL TRIAL: NCT00302289
Title: B181: Stimulation of Thermogenesis by Bio-Active Food Ingredients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Science, Toxicology & Technology, San Francisco, California (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: KF01-188/00
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2000-12

CONDITIONS: Obesity
Keywords: green tea; caffeine; tyrosine; energy expenditure; energy intake
MeSH Terms: conditions — Obesity | interventions — Tyrosine; Tea; Caffeine

INTERVENTIONS:
Drug: tyrosine, green tea, caffeine

SUMMARY:
The primary aim was to measure the effect of green tea extract, tyrosine and caffeine on energy expenditure, appetite ratings and spontaneous energy intake together with recording of side effects in healthy normal weight subjects.

DETAILED DESCRIPTION:
Background: Long-term weight maintenance of a weight loss is often unsuccessful. Often a weight regain is observed in most studies that could indicate that most subjects are not able to change their eating habits. There is a need for simple and safe methods to prevent weight gain and re-gain i.e. by increasing thermogenesis and decrease spontaneous energy intake (EI). Studies have shown that nutritional and food-related non-nutritional factors influence the adjustment of EI and EE as the compounds can enhance the diet-induced thermogenesis (DIT) and suppress appetite.

Method: The present study was designed as a 4-way crossover, randomised, placebo controlled, dou-ble-blind study. Each treatment was separated by >3 d washout period. All treatments were administered as tablets containing either 500 mg green tea extract (whereof 125 mg cate-chins), 400 mg tyrosine, 50 mg anhydrous caffeine, or placebo.

on each test day body weight and composition was assessed. All participants underwent a 4.5-h assessment of energy expenditure by indirect calorimetry in a ventilated hood. Energy intake recorded of an ad libitum pasta salad brunch served after the last hood measurement

Subjects: Twelve healthy lean (20<BMI<25) weight stable non-smoking subjects between 18-40 years of age were tested 4 times each with a wash-out period of at least 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Twelve healthy and normal-weight men (age: 23.72.6 y, BMI: 22.41.8 kg/m2) participated in the study. They were weight stable (within 3-kg in last 3 mo), non-smoking, non-athletic, and had no use of dietary supplements or frequent use of medication.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2000-01; Study Completion 2000-12

PRIMARY OUTCOMES:
heart rate
blood pressure
enegy expenditure
energy intake
subjective appetite sensations

CONTACTS AND LOCATIONS:
Overall Officials: Astrup Arne, Prof, Principal Investigator — Department of Human Nutrition, The Royal Veterinary and Agricultural University, Denmark
Locations (1):
- Department of Human Nutrition, The Royal Veterinary and Agricultural University, Frederiksberg, Denmark